CLINICAL TRIAL: NCT02333097
Title: Prospective Study for Diagnosis Utility of Array-CGH Screening in Case of Non Syndromic Congenital Heart Defect in Prenatal Diagnosis (CAPA)
Brief Title: Non Syndromic Congenital Heart Defect and Array-CGH in Prenatal Diagnosis
Acronym: CAPA
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-A01528-39
Record Dates: First submitted 2014-12-29; First posted 2015-01-07 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Non Syndromic Congenital Heart

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Comparative genomic hybridization (CGH)-based microarrays are now often used during pregnancy in case of fetal polymalformation in order to assess significant genomic alterations. However, it is not clear whether array-CGH provide a diagnostic utility in case of isolated congenital heart defect.

This is the first prospective study aiming at defining the right chromosomal screening when a fetal isolated congenital heart defect is identified by ultrasound.

DETAILED DESCRIPTION:
Comparative genomic hybridization (CGH)-based microarrays are now often used during pregnancy in case of fetal polymalformation in order to assess significant genomic alterations. Up to now, in case of isolated heart defect, only fetal karyotype with FISH 22q11 was usually offered. However, micro deletions or duplications could not be identified elsewhere throughout the genome. Then, in case of fetal chromosomal micro-rearrangements, parents could not be fully informed for global and neurodevelopmental prognosis. To our knowledge, clear-cut study, to assess whether array-CGH provide a diagnostic utility in case of isolated congenital heart defect, don't exist.

After informed consent, 80 women will be enrolled during two years in 2 official prenatal diagnosis centers in France. This survey is assumed to identify at least 8% of unbalanced chromosomal abnormalities. This will be also compared with 22q11 rearrangements rate.

This is the first prospective study aiming at defining the right chromosomal screening when a fetal isolated congenital heart defect is identified by ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman over 18-year-old ;
* Ongoing health insurance ;
* Informed consent ;
* Prenatal samples from amniotic fluid ;
* Isolated congenital heart defect.

Exclusion Criteria:

* Transposition of great arteries ;
* Amniotic fluid sample refusal.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant woman whose a fetal isolated congenital heart defect is identified
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2015-01; Primary Completion 2018-08 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Identification a significant rate of chromosomal imbalances on ACPA > 8% | J0

SECONDARY OUTCOMES:
To compare rates of abnormalities identified by karyotype FISH 22q11 versus ACPA | J0
To compare cardiac ultrasound prenatal data with postnatal data including pathological data (if TOP) | J0
To compare the nature of chromosomal imbalances with the type of MCC | J0

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Pasquier, PH, Principal Investigator — Rennes University Hospital
Locations (2):
- France (2):
  - Rennes University Hospital, Rennes
  - St Brieuc University Hospital, Saint-Brieuc